CLINICAL TRIAL: NCT07122544
Title: The Impact of Pulmonary Rehabilitation Conducted in Therapeutic Salt Chambers on the Clinical Status of Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Pulmonary Rehabilitation in Salt Chambers for Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 169/MN/SD/2025
Record Dates: First submitted 2025-07-30; First posted 2025-08-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-07

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: speleotherapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Breathing Exercises; Relaxation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pulmonary Rehabilitation in Salt Chambers (Experimental): Participants undergo a 16-day pulmonary rehabilitation program conducted in therapeutic salt chambers. The intervention includes general fitness, respiratory and relaxation exercises, health education. Conducted under supervision of a multidisciplinary team (physiotherapist, nurse, dietitian, physician). Sessions take place in the underground salt chambers of the "Wessel" complex (Salt Mine 'Wieliczka', Wieliczka, Poland).
  Interventions: Behavioral: Therapeutic stay in subterranean sanatorium chambers (microclimate therapy); Behavioral: Breathing exercises; Behavioral: General fitness exercises; Behavioral: Relaxation training; Behavioral: Health education
- Surface Rehabilitation (Active Comparator): Participants undergo the same 16-day pulmonary rehabilitation program as in Arm 1, but conducted in standard surface conditions without exposure to salt chamber microclimate.
  Interventions: Behavioral: Breathing exercises; Behavioral: General fitness exercises; Behavioral: Relaxation training; Behavioral: Health education
- Passive Stay in Salt Chambers (Experimental): Participants attend daily 180-minutes passive sessions in therapeutic salt chambers for 16 days, without any physical exercise component.
  Interventions: Behavioral: Therapeutic stay in subterranean sanatorium chambers (microclimate therapy); Behavioral: Health education
- Health education only (Active Comparator): Participants receive printed materials and general health education related to COPD management. No supervised exercise or microclimatic exposure is included.
  Interventions: Behavioral: Health education

INTERVENTIONS:
Behavioral: Therapeutic stay in subterranean sanatorium chambers (microclimate therapy) — Characteristics of the underground environment in the Wieliczka sanatorium chambers:
  Stable climatic conditions: relative humidity ranging from 60-75%, temperature between 12.9-14.5°C; High chemical and biological air purity; Mineral content in the air: 2.7-8.1 mg/m³, consisting mainly of chloride, sodium, potassium, calcium, and fluoride ions; Air ionization: 1,200-4,700 aeroions/cm³ of air. Elevated atmospheric pressure: increased by approximately 16-20 mmHg compared to surface conditions.
  Arms: Passive Stay in Salt Chambers; Pulmonary Rehabilitation in Salt Chambers
Behavioral: Breathing exercises — 30 minutes daily. Breathing exercises will include active respiratory exercises, drainage and effective coughing techniques, resistance training of the respiratory muscles, chest mobilization and relaxation exercises, breathing through pursed lips, as well as short and prolonged exhalation exercises.
  Arms: Pulmonary Rehabilitation in Salt Chambers; Surface Rehabilitation
Behavioral: General fitness exercises — 30 minutes daily. General conditioning exercises will incorporate components aimed at improving overall aerobic capacity (e.g., walking-based activities, dance routines, step exercises), flexibility and coordination (e.g., stretching and balance exercises), and strength (e.g., exercises using resistance bands or dumbbells). The training will be conducted in interval, circuit, and free-form formats. Resistance levels will be individually adjusted to the patient's capacity.
  Arms: Pulmonary Rehabilitation in Salt Chambers; Surface Rehabilitation
Behavioral: Relaxation training — 30 minutes, once during the entire cycle. Relaxation training will include rest in a seated position, with dimmed lighting and calming music.
  Arms: Pulmonary Rehabilitation in Salt Chambers; Surface Rehabilitation
Behavioral: Health education — Educational materials in printed form for distribution covering the following topics:
  COPD - information about the disease;
  Breathing exercises and bronchial hygiene;
  Benefits of physical activity, including examples of exercises that can be performed at home.

SUMMARY:
Title: The Impact of Pulmonary Rehabilitation Conducted in Therapeutic Salt Chambers on the Clinical Condition of Patients with Chronic Obstructive Pulmonary Disease

Background and Rationale:

Chronic Obstructive Pulmonary Disease (COPD) is a progressive respiratory disorder that significantly reduces patients' quality of life and functional capacity. In the search for supportive therapeutic strategies, there is growing interest in unconventional therapeutic environments such as therapeutic salt chambers. The underground climate of the "Wieliczka" Salt Mine in Poland - characterized by humidity 60-75%, temperature 12.9-14.5°C, high air purity and ionization - has shown therapeutic potential. However, the clinical effects of pulmonary rehabilitation conducted in such an environment in COPD patients remain insufficiently documented.

Study Objective:

To evaluate the effect of pulmonary rehabilitation and climatic therapy conducted in underground salt chambers on the clinical condition of patients with stable COPD.

Research Question:

Does pulmonary rehabilitation conducted in a subterranean salt mine environment offer measurable clinical benefits compared to standard surface-based rehabilitation?

Study Design and Methods:

This is a randomized, controlled, four-arm interventional study including 80 adult patients with a confirmed diagnosis of COPD according to the GOLD 2025 criteria. Participants will be randomly assigned to one of four groups:

Group A: Pulmonary rehabilitation in underground therapeutic salt chambers (physical training + microclimate exposure).

Group B: Pulmonary rehabilitation in a surface-level gymnasium (physical training without microclimate exposure).

Group C: Passive stay in underground salt chambers (microclimate exposure without physical training).

Group D: Health education only (control group, surface level).

The intervention program consists of 16 consecutive working days of 3-hour daily sessions. The content of the rehabilitation varies depending on the assigned group and includes general conditioning exercises, respiratory exercises, relaxation training, and health education.

Outcome Measures and Assessment Tools:

Clinical assessments will be conducted at three time points: prior to the intervention (T0), immediately after the intervention (T1), and at a 3-month follow-up (T2 - for Groups A and B only). The monitored variables include:

Exercise Tolerance: Incremental Shuttle Walk Test (ISWT)

Health-Related Quality of Life: St. George's Respiratory Questionnaire

COPD Symptoms and Risk Indexes: COPD Assessment Test (CAT), BODE Index

Muscle Strength: Deadlift test, hand dynamometer, 30-second Chair Stand Test

Respiratory Muscle Strength: Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP)

Body Composition: Bioelectrical Impedance Analysis (BIA)

Dyspnea Scales: Borg Scale, modified Medical Research Council (mMRC) scale

Chest Mobility: Measuring tape assessment

The study is designed to evaluate both the immediate and long-term effects of different pulmonary rehabilitation models on clinical outcomes in COPD patients, with a focus on whether the underground environment enhances rehabilitation efficacy.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis confirmed by a pulmonology specialist according to the 2025 GOLD guidelines.
* FEV1 ≥ 30% of the predicted value.
* FEV1/FVC < 0.7 after bronchodilator administration in spirometry.
* Negative bronchodilator reversibility test.
* Voluntary written consent to participate in the study.

Exclusion Criteria:

* COPD exacerbation.
* Active cancer or a history of cancer within the past five years.
* Musculoskeletal disorders preventing independent movement and participation in exercise tests and training included in the study protocol.
* Recent (within six months) surgical procedure or trauma to the chest, abdomen, skull, brain, or eye area.
* Severe valvular heart disease.
* Implanted cardioverter-defibrillator.
* Diagnosed arrhythmias posing a risk of loss of consciousness.
* Acute coronary artery disease.
* Epilepsy.
* Uncontrolled arterial hypertension despite medication.
* Primary or secondary immunodeficiencies.
* Respiratory failure requiring chronic or intermittent oxygen therapy.
* Infectious diseases with fever during the experiment or within two weeks before the study.
* Claustrophobia.
* Pregnancy.
* Simultaneous participation in another rehabilitation program.
* Significant changes in pharmacological treatment during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in exercise tolerance (ISWT distance) | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Incremental Shuttle Walk Test (ISWT) used to assess functional exercise tolerance in COPD patients. Measured as distance walked in meters. Evaluates change from baseline to post-intervention and at 3-month follow-up to assess immediate and sustained effects of rehabilitation.
Change in quality of life (SGRQ-C total score) | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  St. George's Respiratory Questionnaire version COPD (SGRQ-C) measures disease-specific quality of life.

SECONDARY OUTCOMES:
Change in Respiratory Muscle Strength | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Respiratory Muscle Strength: Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP)
Change in Chest Mobility | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Measured using thoracic expansion assessment during respiration.
Change in COPD Symptoms Severity | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Evaluated using the COPD Assessment Test (CAT).
Change in Dyspnea Severity | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Measured using the Modified Medical Research Council (mMRC) Dyspnea Scale and Borg Dyspnea Scale.
Change in Muscle Strength | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Assessed with the 30-Second Chair Stand Test (30sCST), handgrip dynamometry, and deadlift strength test.
Thigh circumference | Baseline (Day 1), Post-intervention (Day 18), 3 months follow-up (Day 108)
  Circumferential measurement of both thighs at their widest point with a tailor's tape measure.

OTHER OUTCOMES:
BODE Index | Baseline (Day 1 only)
  Multidimensional index including BMI, airflow obstruction (FEV1), dyspnea (mMRC), and exercise capacity (the result of the Incremental Shuttle Walk Test (ISWT) will be converted to an estimated equivalent distance of the 6-Minute Walk Test (6MWT) using established predictive formulas). In this study, the BODE index will be calculated only at baseline using data collected on Day 1. It will not be reassessed during follow-up visits because spirometry (FEV₁ measurement) will not be repeated after baseline.
Post-Bronchodilator Spirometry | Baseline (Day 1 only)
  A single spirometry with bronchodilator reversibility testing will be performed at baseline according to American Thoracic Society (ATS) and European Respiratory Society (ERS) standards. Spirometry will be performed only once during the study and will not be repeated at any subsequent visits.
  Parameters recorded:
  FEV₁ (Forced Expiratory Volume in 1 second) - liters and % predicted FVC (Forced Vital Capacity) - liters and % predicted FEV₁/FVC ratio
  Post-bronchodilator values will be used exclusively for participant eligibility assessment according to GOLD 2025 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- AKF Kraków, Krakow, Małopolska, Poland